CLINICAL TRIAL: NCT07356739
Title: Phoenixin-14 Downregulation as a Novel Prognostic Biomarker in Sepsis: Molecular and Clinical Evidence
Brief Title: Phoenixin-14 Downregulation in Sepsis
Status: Completed | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gulsum Altuntas, Doctor, Firat University
Other Study IDs: 23376
Record Dates: First submitted 2025-08-15; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sepsis - to Reduce Mortality in the Intensive Care Unit; Sepsis Biomarker; Phoenixin-14 Molecular Downregulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Sepsis is a leading cause of morbidity and mortality in intensive care units (ICUs) worldwide, accounting for millions of deaths annually. Despite the use of established biomarkers such as procalcitonin, C-reactive protein (CRP), and interleukin-6 (IL-6), their predictive accuracy for mortality remains suboptimal. Phoenixin-14 (PNX-14), a neuropeptide with demonstrated anti-inflammatory and antioxidant effects in preclinical studies, has not been extensively investigated in the context of sepsis. This study aimed to evaluate the prognostic value of serum PNX-14 levels and gene expression in predicting hospital mortality among ICU patients with sepsis.

Methods:

This prospective observational cohort study included 77 adult patients admitted to a tertiary ICU with a diagnosis of septic shock between March and November 2024. Patients under 18 years, pregnant women, and those with chronic steroid use, immunosuppression, malignancy, severe liver disease, or early discharge/death within 72 hours of diagnosis were excluded. Upon ICU admission, demographic and clinical data were recorded, including Acute Physiology and Chronic Health Evaluation II (APACHE II) and Sequential Organ Failure Assessment (SOFA) scores. Serum PNX-14, CRP, procalcitonin, IL-1β, IL-6, tumor necrosis factor-α (TNF-α), and IL-10 levels were measured using ELISA. Gene expression levels of PNX-14 were quantified via real-time PCR. The primary endpoint was hospital mortality; secondary endpoints included associations and correlations between PNX-14 levels, inflammatory markers, and severity scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 admitted to our tertiary intensive care unit with diagnoses of sepsis and/or septic shock

Exclusion Criteria:

* Patients under the age of 18, patients who were discharged/transferred or died within 72 hours after being diagnosed with sepsis, patients/relatives who refused to participate in the study, pregnant women, patients with chronic steroid use, endocrinopathy, liver disease, malignancy, or a history of immunosuppression.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 admitted to our tertiary intensive care unit with diagnoses of sepsis and/or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
The association between PNX14 levels (serum ELISA) and intensive care mortality in patients with sepsis/septic shock | Blood samples were collected within 2 hours of ICU admission, mortality is taken through study completion, an average of 1 year.
  EEndpoints: to evaluate supression of PNX-14 (serum ELISA) at the molecular level in patients with sepsis and their potential as a translational biomarker. The correlation between PNX14 levels and those of CRP, procalcitonin, IL-1β, IL-6, IL-10, and TNF-α levels were also examined (serum ELISA) as part of the endpoints.
the relationship between PNX14 levels and in-hospital mortality in patients with sepsis or septic shock | within 2 hours of ICU admission

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT07356739/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT07356739/ICF_001.pdf